CLINICAL TRIAL: NCT04244292
Title: Evaluation of the Accuracy and Reliability of the Percentage of Glottic Opening Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Assoc Prof, Diskapi Teaching and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: POGO Score
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-01

CONDITIONS: Intubation
Keywords: Intubation; Laryngeal view; Scoring systems; Larynx
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Videolaryngoscopy (Other): Patient will be intubated by using videolaryngoscope
  Interventions: Other: Videolaryngoscopy

INTERVENTIONS:
Other: Videolaryngoscopy — Patient will be intubated by using videolaryngoscope

SUMMARY:
Current classifications of the laryngeal view during laryngoscopy are criticized for being subjective.

The modified CL classification is criticized as it does not predict difficult intubation and especially grade 2 is operator dependent and partial view is not well defined. The numerical expression of the percentage of the glottic aperture (POGO = percentile of glottic opening) is another score. In this score, A POGO score of 100% accounts for full visualization of the larynx starting from anterior commissure to the posterior cartilage, while 0% indicated a complete absence of glottic opening. Previous validation studies reported on the reliability of POGO; however, accuracy was not evaluated.

The use of a standard and effective classification method will facilitate and accelerate communication between anesthetists in difficult life-threatening situations such as difficult airway / difficult intubation / difficult ventilation and contribute to patient safety. The use of common terminology can also facilitate the evaluation of the performance of intubation tools. The aim of this study was to evaluate the accuracy and intra and inter rater reliability of the POGO score

DETAILED DESCRIPTION:
Reviewer anesthesiologist will be asked to score still images of laryngeal views, which will be obtained from patients requiring intubation for general anesthesia, after obtaining written informed consent. The images of the larynx will be captured first with the Macintosh blade and thereafter with the D blade. An expert panel will score these images with the Cormack Lehane and POGO scores. The set of images will be prepared from patients with both difficult and normal airway anatomy. Some images in the series will be repeated to assess intra rater variability. The anesthesiologist will be asked to rate 20 images both with the CL and POGO scores. The experience of the raters in airway management, their experience with videolaryngoscopy and scoring systems used currently when documenting videolaryngoscopy and demographic data will be also obtained. The POGO scores of the participants and investigators will be compared. The primary outcome measure was the reviewer's agreement with the correct POGO scores (accuracy).

ELIGIBILITY:
Inclusion Criteria:

• Patients receiving general anesthesia

Exclusion Criteria:

• Emergency surgery-

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Percentile of glottic opening | 2 minutes after induction of anesthesia
  A percentile of glottic opening score of 100% accounts for full visualization of the larynx starting from anterior commissure to the posterior cartilage, while 0% indicated a complete absence of glottic opening.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Unal, Principal Investigator — UNIVERSITY OF HEALTH SCIENCES DISKAPI YILDIRIM BEYAZIT TEACHING HOSPITAL
Locations (1):
- Ankara Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norris A, Heidegger T. Limitations of videolaryngoscopy. Br J Anaesth. 2016 Aug;117(2):148-50. doi: 10.1093/bja/aew122. Epub 2016 Jun 1. No abstract available. PMID 27251753
- [Background] Ochroch EA, Hollander JE, Kush S, Shofer FS, Levitan RM. Assessment of laryngeal view: percentage of glottic opening score vs Cormack and Lehane grading. Can J Anaesth. 1999 Oct;46(10):987-90. doi: 10.1007/BF03013137. PMID 10522589
- [Background] Cook TM. A grading system for direct laryngoscopy. Anaesthesia. 1999 May;54(5):496-7. doi: 10.1046/j.1365-2044.1999.0907f.x. No abstract available. PMID 10995154